CLINICAL TRIAL: NCT04298970
Title: Novel Organic Kale Products for Prevention of Obesity/Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Future Food Innovation (Industry)
Responsible Party: Principal Investigator, Per Bendix Jeppesen, Associate. Prof, Phd, Diabetes and hormone diseases, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AU/AUH
Record Dates: First submitted 2020-03-03; First posted 2020-03-06 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Consuming a product containing 35-40 gram of freeze dried kale a day.
  Interventions: Dietary Supplement: Intervention
- Placebo (Placebo Comparator): Consuming a placebo product.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Intervention — Freeze-dried Brassica oleracea var. acephala
  Arms: Intervention
Dietary Supplement: Placebo — Placebo product
  Arms: Placebo

SUMMARY:
Investigating the health beneficial effects of freeze-dried Brassica oleracea var. acephala with a high content of fibers, protein, vitamin, minerals, and secondary metabolites on patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, dietary treatment and/or with oral anti-diabetics
* Diabetes debut > 30 year
* Plasma fasting blood glucose > 4mM and < 12 mM
* HbA1c > 43 and ≤ 108 mmol/mol
* BMI between 23-40 kg/m2
* Fasting triglyceride > 1.7 mmol/L and HDL-cholesterol, men: < 1.03 mmol/L and women: 1.29 mmol/L.

Exclusion Criteria:

* Participating or have been participating in other clinical trials within the last 2 months.
* In treatment with insulin, systemic glucocorticoids, glitazones or GLP-1 analogs.
* Cardiovascular-, physiological-, neurological-, and/or kidney diseases.
* Alcohol- or pill abuse.
* Acute diseases.
* Blood pressure ≥ 160/100
* Pregnant or breastfeeding women.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
iAUC | Throughout the study (up to 1 year)
  The blood glucose incremental area under curve, OGTT

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No